CLINICAL TRIAL: NCT01686464
Title: A New Clinical Therapy for Bell's Palsy
Brief Title: A Clinical Study on the Combined Magnetic and Oxygen Treatment for Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, wang yanliang, principal investigator, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: wykq2012; 665533 (Other: WZMC)
Record Dates: First submitted 2012-08-28; First posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Bell's Palsy
Keywords: magnetic; oxygen; Bell's Palsy; acupuncture
MeSH Terms: conditions — Bell Palsy | interventions — Prednisone; Valacyclovir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnetic - Oxygen (Experimental): Magnetic and Oxygen Treatment for Bell's Palsy
  Interventions: Device: Magnetic and Oxygen Treatment
- prednisone - valacyclovir (Active Comparator): prednisone and valacyclovir treatments for bell palsy
  Interventions: Drug: prednisone and valacyclovir treatments

INTERVENTIONS:
Drug: prednisone and valacyclovir treatments — patients were administered prednisone as a single dose of 40 mg daily for 5 days; the dose will then be reduced by 10 mg per 5 day, with a total treatment time of 20 days.while taking valacyclovir 400 mg in three doses daily for 10 days.
  Other Names: prednisone and valacyclovir
  Arms: prednisone - valacyclovir
Device: Magnetic and Oxygen Treatment — MOMC treatment was given as daily 20 min section for 10 days with 2~3 days of intermission between. Oxygen therapy was given simultaneously at a flow rate of 2~3.0 L / min for the same duration during all acupuncture sections.
  Arms: Magnetic - Oxygen

SUMMARY:
The aim of this clinic trial is to testify the efficacy of using new and noninvasive therapy, called simultaneous "Magnetic and Oxygen Treatment along Meridians and Collaterals" (MOMC), to treat Bell's Palsy.

DETAILED DESCRIPTION:
Between June 1998 and January 2005, a total of 3002 subjects with BP were evaluated, 882 patients fulfilled the inclusion criteria and entered the study.

Patients were randomly assigned to either the prednisone-valacyclovir group(group 1) or the magnetic-oxygen group(group 2) . Among the 882 patients completing the study,825 patients in group 1 received prednisone, given as a single dose of 40 mg daily for 5 days; the dose will then be reduced by 10 mg per 5 day, with a total treatment time of 20 days.while taking valacyclovir 400 mg in three doses daily for 10 days. 57 patients in group 2 received magnetic-oxygen treatment:MOMC treatment was given as daily 20 min section for 10 days with 2~3 days of intermission between;Oxygen therapy was given simultaneously at a flow rate of 2~3.0 L / min for the same duration during all acupuncture sections.

Clinical evaluation for the severity of paralysis was performed immediately before and after the treatment using the facial nerve grading (FNG) scores of House and Brackmann system.

ELIGIBILITY:
Inclusion Criteria:

1. Only patients with complete (or nearly complete) non-recurrent facial paralysis (grade 5-6/6) for more than 1 months
2. the first time to onset the disease
3. on one side of the face paralysis
4. willing to finish the whole observation period
5. with written consent form signed by themselves.

Exclusion Criteria:

1. facial palsy caused by other disease, such as infectivity multiple radiculitis, tumor which offend temporal bone, cerebral trauma
2. facial palsy combine diabetes, the severe disease of heart vessel, cerebral vessel, liver, kidney, lung, and psychosis
3. patient with Hunt's syndrome
4. pregnant women or women in lactation
5. patients are participating other clinical research

Ages: 10 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 1998-06; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
House-Brackmann scale | the 20th day of completion of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: yan L wang, Ph .D, Principal Investigator — Wenzhou Medical University; Ping Li, M.D., Study Chair — The 4th military medical university
Locations (1):
- the 4th Military Medical University, Xi’an, Shanxi, China

REFERENCES:
- [Result] Shafshak TS, Essa AY, Bakey FA. The possible contributing factors for the success of steroid therapy in Bell's palsy: a clinical and electrophysiological study. J Laryngol Otol. 1994 Nov;108(11):940-3. doi: 10.1017/s0022215100128580. PMID 7829945
- [Result] Finsterer J. Management of peripheral facial nerve palsy. Eur Arch Otorhinolaryngol. 2008 Jul;265(7):743-52. doi: 10.1007/s00405-008-0646-4. Epub 2008 Mar 27. PMID 18368417
- See also: Bell palsy paralysis Acupuncture — http://www.nlm.nih.gov/medlineplus/bellspalsy.html